CLINICAL TRIAL: NCT03679325
Title: Heart Rate Variability in Healthy Older and Older COPD After Vitamine D Use and Whole Body Vibration Protocol
Brief Title: Evaluation of Cardiac Variability After a Vitamine D Protocol and Whole Body Vibration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maíra F Pessoa (Other)
Responsible Party: Sponsor-Investigator, Maíra F Pessoa, Clinical Professor, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: COPDcardiac variability
Record Dates: First submitted 2018-09-19; First posted 2018-09-20 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Copd; Aging
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitamine D (Active Comparator): a dose once a week
  Interventions: Dietary Supplement: vitamine D; Other: whole body vibration (WBV)
- vitamine D placebo (Placebo Comparator): a dose once a week
  Interventions: Other: whole body vibration (WBV)

INTERVENTIONS:
Dietary Supplement: vitamine D — a dose once a week
  Arms: vitamine D
Other: whole body vibration (WBV) — 03 months of WBV training three times per week

SUMMARY:
Evaluation of heart rate variability in time and frequency domains, in Chronic Obstructive Pulmonary Disease (COPD) after 03 months of vitamine D supplementation and whole body vibration (WBV) training

ELIGIBILITY:
Inclusion Criteria:

* COPD or healthy elderly sedentary according to International Physical Activity Questionnaire
* BMI between 22.9 and 28 kg/m2
* COPD with clinical-functional diagnosis of the disease according to Gold
* ex-smokers

Exclusion Criteria:

* Older patients with COPD who had episodes of exacerbation in the last three months
* Who participate in pulmonary rehabilitation programs in the last year
* Who used home oxygen therapy
* Patients with COPD-associated comorbidities
* Who were taking vitamin D

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
heart rate variability | before and immediately after the chronic intervention
  evaluation of time and frequency domains

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Williamson A, Martineau AR, Jolliffe D, Sheikh A, Janssens W, Sluyter J, Rafiq R, de Jongh R, Griffiths CJ. Vitamin D for the management of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2024 Sep 27;9(9):CD013284. doi: 10.1002/14651858.CD013284.pub2. PMID 39329240